CLINICAL TRIAL: NCT02044978
Title: Initial Fixation of Bisphosphonate-coated Dental Implants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Per Aspenberg (Other)
Responsible Party: Sponsor-Investigator, Per Aspenberg, professor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tandskruv tidsserie
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Pre-integration Failure of Dental Implant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bisphosphonate implant (Active Comparator): Dental implant coated with zoledronate Note: Both arms in each patient (2 implants)
  Interventions: Device: Zoledronate-coated dental implant
- control (Placebo Comparator): Dental implant without coating Note: Both arms in each patient (2 implants)

INTERVENTIONS:
Device: Zoledronate-coated dental implant
  Arms: Bisphosphonate implant

SUMMARY:
16 patients will be included. Each patient receives 2 dental implants. One of them is coated with a drug, zoledronate, to improve fixation. Fixation is measured by vibration resonance frequency analysis at insertion and 2, 4, 6 and 8 weeks after insertion.The 2 implants in each patient are compared. We expect to find an early improvement (higher resonance frequency) in the coated implant.

DETAILED DESCRIPTION:
The zoledronate is linked to the titanium implant surface via a nanolayer of crosslinked fibrinigen. Resonance frequency is measured with standard clinical equipment (Ostell apparatus).

ELIGIBILITY:
Inclusion Criteria:

Need for dental implant in upper jaw. CTscan showing at least 6 mm bucco-lingual thickness. Generally healthy

Exclusion Criteria:

Drugs or conditions that influence or are thought to influence bone healing, such as bisphosphonates, corticosteroids, other oral pathologies, severe autoimmune diseases, cancer. Osteoporosis is not cause for exclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Vibration frequency ratio | 4 and 6 weeks
  Each patients has a study implant and a control implant. Their change vibation frequency from insertion till measurement time point is measured and the ratio between changes for the 2 implants forms the outcome measure. Avarage values for 4 and 6 weeks will be used.

SECONDARY OUTCOMES:
Marginal resorption | 8 weeks
  Radiographic loss of bone at the margin of the implant, measured as difference in mm from the superficial bone contour between insertion and 8 weeks.
Vibration: area under the curve | 2-8 weeks
  Each patients has a study implant and a control implant. Their change vibation frequency from insertion till measurement time point is measured and the ratio between changes for the 2 implants forms the outcome measure. Avarage values for all weeks will be used.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Käkcentralen, Linköping
  - Tandläkarhuset, Linköping